CLINICAL TRIAL: NCT04056546
Title: Interest of Rapid Typing in Adenovirus Infections: Sensitivity and Specificity, Study of the Association Clinical Characteristics and Viral Type.
Brief Title: Interest of Rapid Typing in Adenovirus Infections.
Acronym: TYPADENO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2011/08
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Adenovirus; Adenovirus Disease; Genotyping
Keywords: Real-time Polymerase-Chain Reaction
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biological samples identified as Adenovirus positive (Hexon quantitative PCR positive samples) by the University Hospital's Virology laboratory, carried out for diagnostic purposes since January 2008, and stored at -80 ° C.
Oversight: Data Monitoring Committee: No

SUMMARY:
Proposal of a "rapid typing" technique by a new real-time PCR method, simpler, faster and cheaper than nucleotide sequencing (reference method) for rapid typing in Adenovirus infections.

DETAILED DESCRIPTION:
Adenoviruses cause many infections, mainly respiratory and gastroenteric, in pediatrics.

They also behave as opportunistic agents in 10% of hematopoietic stem cell recipients. In these immunocompromised persons, these infections are all the more frequent as the graft is of placental origin and the recipient a child (20%). They are then willingly disseminated and potentially deadly; their treatment is based on cidofovir, a viral agent that is very sensitive to handling.

Adenoviruses, which have a high genetic diversity, are classified into 7 types. According to some observations, still limited, some types of Adenovirus would show a higher pathogenicity (types C and A). Thus, viral typing may be prognostic for immunocompromised patients, justifying the initiation of an earlier specific treatment when identifying certain more pathogenic viral types, in addition to measuring the viral load, already performed by quantitative PCR.

For this purpose, this study proposes a "fast typing" technique by new real-time PCR method, simpler, faster and cheaper than nucleotide sequencing, reference method.

ELIGIBILITY:
Inclusion criteria:

- viral load greater than or equal to 10 ^ 4 copies / mL (blood and body fluids) or copies / gram of stool or copies / μg of DNA (biopsies).

Exclusion Criteria:

* Samples identified as positive in Adenovirus, not re-analyzable (insufficient sample quantity, alteration during thawing).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Therefore inclusion in this study of any patient having at least a viral load greater than or equal to 10 ^ 4 copies / mL (blood and body fluids) or copies / gram of stool or copies / μg of DNA (biopsies) for the duration study.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2014-07-04 (Actual); Study Completion 2014-07-04 (Actual)

PRIMARY OUTCOMES:
Type viral characterization (scale A to G) | At the screening
  sensitivity and specificity of the rapid typing technique, expressed for each strain, relative to the reference method (nucleotide sequencing), among initial diagnostic samples of viral load> 10 ^ 4 / mL.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Edith LAFON, Pr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No